CLINICAL TRIAL: NCT00234715
Title: A Pilot Study: Psychosocial and Socio-Demographic Determinants of Accepting Breast Cancer Risk Assessment
Brief Title: Psychosocial Study on Breast Cancer Risk Assessment
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Other Study IDs: UHNREB#05-0601-CE
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2007-11-15 (Estimated); Status verified 2007-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast Cancer Risk; Breast Cancer Risk Assessment; Psychosocial; Acceptance
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The proposed pilot study is part of the design and development process of a final questionnaire that aims to gain insight on factors that influences acceptance and adoption of breast cancer risk assessment in women. Feedback on the questionnaire will help identify potential issues of clarity, comprehensibility, and reliability; and to identify possible biases that often accompany a designed questionnaire. Information gained from the large-scale study will provide directions for the development of educational strategies in the TIBS research program that could accompany increases in public awareness of risk factors, the availability of risk assessment tools and preventive lifestyle.

DETAILED DESCRIPTION:
The development of risk assessment tools for preventive oncology aims to identify all members of a given at risk subpopulation to whom intervention strategies can be offered to reduce their risk. An ideal risk assessment tool should permit assessment of a woman's breast cancer risk in order to a) identify the needs for and potential benefits of risk reducing interventions; b) direct her to the most appropriate risk reducing interventions, and; c) monitor the efficacy of the intervention in actually reducing risk. Earlier implemented risk reduction interventions could potentially preclude needs for more drastic lifestyle and less desirable changes, such as chemoprevention and prophylactic surgeries, later in life. Currently, no such classification and monitoring technique has proven effective. Yet several candidate techniques are being investigated. While risk assessment tools may potentially provide future benefits, the effectiveness of current and new risk assessment tool developments certainly requires users to perceive these tools as potentially effective. It is this perception of potential effectiveness that would motivate them to adhere to risk assessment protocols the evaluation of which would help provide the evidence base for understanding true effectiveness. The investigators of this study are currently developing a Transillumination Breast Spectroscopy (TIBS) research program, consisting of ongoing studies of different types. As part of the technology assessment process for TIBS, and in part due to the further development of the research program, there is a need to address factors that may directly or indirectly influence willingness to participate in a breast cancer risk assessment. The primary goal of this pilot study is to determine the content validity of the investigator-designed draft questionnaire. The outcome measure of a final questionnaire is to assess general acceptability of breast cancer risk assessment and degree of acceptability based on a) knowledge and awareness of breast cancer, b) varying levels of involvement and invasiveness of a risk assessment procedure, and c) perceived potential effectiveness of risk reducing interventions. Acceptability of risk assessment, willingness to undergo therapy and follow through with recommendations is assessed independent of currently available and new developments of risk assessment procedures.The secondary goal of this study is to test the overall comprehensibility (e.g. language, clarity), question acceptability (e.g. appropriateness of response selection), and reliability of the questionnaire.Information gained from this pilot study will be considered in the development of a final questionnaire to be administered to a large population representative cohort. The results of the planned future study will provide directions for the development of educational strategies in the TIBS research program that should accompany increases in public awareness on risk factors, the availability of risk assessment tools and preventive lifestyle and insight into the extent of broad-based community education strategies required to initiate and sustain interest in assessment for breast cancer risk among women in the general public to facilitate informed decision-making related to breast health in these women. Critical gaps in knowledge of risk factors and preventive lifestyle changes identified in this subsequent study can provide a focus for the educational strategies, which may address: the costs of risk assessment (e.g. stress, financial, inconvenience) and the development of understandable and practical educational materials to ensure their accessibility to a broad range of audiences, including those women who may be candidates for risk reducing interventions but who are not yet aware of its availability. The ultimate hypothesis of a future large-scale study is:General knowledge and awareness of breast cancer, psychosocial factors such as perceived risk susceptibility and perceived costs of risk assessment (e.g. stress, financial, inconvenience), perceived effectiveness of intervention strategies, and socio-demographic position are determinants of accepting risk assessment.However, to help guide questionnaire design and development, a pilot study is required to identify issues of the questionnaire such as content validity, overall comprehensibility (e.g. language, clarity), question acceptability (e.g. appropriateness of response selection), and reliability. To achieve the goals of the pilot study, we intend to recruit 50 women between ages of 25 - 74 years (10 per age group, 25 - 34, 35 - 44, 45 - 54, 55 - 65, 65 - 74). A 26-item investigator-designed, self-administered questionnaire was designed with standard measures. The questionnaire consists of 7 sections covering the following topics: Breast Cancer Knowledge and Awareness, Susceptibility Perception, Likelihood of Undergoing Risk Assessment, Benefits and Barriers of Risk Assessment, Breast Cancer Risk Assessment, Risk Reduction Intervention, and Demographics

ELIGIBILITY:
Inclusion Criteria:

* Are 25 - 74 years of age
* Are in good health

Ages: 25 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort recruited from the University Health Network community.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2005-10; Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lothar Lilge, PhD, Principal Investigator — Ontario Cancer Institute, University Health Network, Toronto, Ontario, Canada M5G 2M9; Department of Biophysics and Bioimaging, University of Toronto, Toronto, Ontario, Canada M5G 2M9
Locations (1):
- Ontario Cancer Institute / Princess Margaret Hospital, Toronto, Ontario, Canada